CLINICAL TRIAL: NCT03832166
Title: A Prospective, Randomized Two Group Study to Evaluate the Feasibility and Initial Efficacy of a Community-engaged Screening, Identification, and F&V Intervention to Improve F&V Intake and CKD Outcomes in 140 AA Adults
Brief Title: Reducing Chronic Kidney Disease Burden in an Underserved Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R21DK113440-01A1 (NIH)
Record Dates: First submitted 2019-02-01; First posted 2019-02-06 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-07

CONDITIONS: CKD; ESRD
Keywords: CKD; Low Income; Diet; Fruits and Vegetables
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Fruit; Vegetables; Cooking

STUDY DESIGN:
Intervention Model Description: Prospective, randomized two group study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fruits and Vegetables Only (Experimental): This group will receive a prescribed amount of free fruits and vegetables (F & V) for 6 weeks through pick-up at a farm stand, or direct delivery. After 6 weekly pick-up/deliveries, participants will be provided vouchers and reminders to obtain F&V at farm stands for an additional 18 weeks with minimal contact
  Interventions: Other: Fruits and Vegetables
- Fruits and Vegetables and Cook (Experimental): In addition to the prescribed amount of free F&V, participants will receive 6 weekly, group nutrition and cooking education classes based on "The Happy Kitchen" curriculum. Participants will also receive free ingredients to complete the recipe from each weekly session at home.
  Interventions: Other: Fruits and Vegetables; Other: Cooking

INTERVENTIONS:
Other: Fruits and Vegetables — Fruits and vegetables delivery, once/week for 24 weeks
Other: Cooking — Nutrition education and cooking instruction class, one class/week for 6 weeks
  Other Names: The Happy Kitchen
  Arms: Fruits and Vegetables and Cook

SUMMARY:
To evaluate a scalable population health strategy to 1) screen, 2) identify, and 3) intervene with individuals at high risk of CKD progression to ESRD that could be implemented in other high risk communities and health care systems. This novel study will evaluate the feasibility and preliminary efficacy of providing F&V to individuals identified at high risk study for CKD and ESRD through community health screenings. Further, it will evaluate whether providing education as to how to prepare F&V for consumption, the latter being done for all F&V recipients in PI's preliminary published studies but its efficacy was not specifically tested, increases F&V intake and thereby reduces CKD progression risk as well as related clinical outcomes.

DETAILED DESCRIPTION:
"Fruits and Veggies for Health" is a prospective, randomized two group study to evaluate a community-engaged screening, identification, and F&V intervention to improve CKD outcomes in 140 AA adults (greater than 18 years). Participants will be randomized to a 1) F&V only (F&V Only), or 2) F&V plus a nutrition/cooking program (F&V + Cook).

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate in 6 month F&V study
* Positive urine dipstick.
* African American (self declared) race
* Access to internet via personal computer or mobile device
* Ability to read and write in English

Exclusion Criteria:

* Negative urine dipstick
* Currently receiving dialysis or needing dialysis (stage 5 Kidney disease)
* Have received or need kidney transplant
* Pregnant or plan to become pregnant in the next 6 months
* Baseline urine potassium > 60 mEq/g creatinine
* Nephrotic proteinuria demonstrated on urine ACR measurement
* Lacking access to the internet via personal computer or mobile device
* Unable to read or write in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2020-06-13 (Actual); Study Completion 2020-07-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline concentration of Urine angiotensinogen (AGT) at 6 weeks and 6 months | Baseline; 6 weeks; 6 months
  Primary surrogate marker of eGFR
Change from baseline of Urine albumin-to-creatinine ratio (ACR) at 6 weeks and 6 months | Baseline; 6 weeks; 6 months
  Measure of renal damage
Changes from baseline in fruit and vegetable intake at 6 weeks and 6 months | Baseline; 6 weeks; 6 months
  Track changes in fruit and vegetable intake via ASA24 food diary
Changes from baseline in dietary fat intake at 6 weeks and 6 months | Baseline; 6 weeks; 6 months
  Track changes in fat (g) intake via ASA24 food diary
Changes from baseline in caloric intake at 6 weeks and 6 months | Baseline; 6 weeks; 6 months
  Track changes in total caloric(kcal) intake via ASA24 food diary

SECONDARY OUTCOMES:
Changes from baseline in systolic and diastolic Blood pressure at 6 weeks and 6 months | Baseline; 6 weeks; 6 months
  Measure changes in systolic/diastolic blood pressure (mm Hg) to assess cardiovascular disease risk (CVD)
Changes from baseline in serum Lipoprotein levels at 6 weeks and 6 months | Baseline; 6 weeks; 6 months
  Measure changes in total cholesterol, HDL, and LDL (mg/dL) by fingerstick to assess CVD risk
Changes from baseline in serum Glycosolated hemoglobin A1C (HgA1C) levels at 6 weeks and 6 months | Baseline; 6 weeks; 6 months
  Measure changes in HgA1C (mg/dL) by fingerstick as a marker of diabetes and to assess CVD risk
Changes from baseline in Blood glucose at 6 weeks and 6 months | Baseline; 6 weeks; 6 months
  Measure fasting glucose(mg/dL) as a marker of diabetes and to assess CVD risk
Changes from baseline in Body mass index (BMI) at 6 weeks and 6 months | Baseline; 6 weeks; 6 months
  Measure body mass index(lb/inches squared) to assess CVD risk

CONTACTS AND LOCATIONS:
Overall Officials: Donald Wesson, MD, MBA, Principal Investigator — Baylor RI
Locations (1):
- Baylor Research Institute, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available within 6 mths of outcome publication

REFERENCES:
- [Background] Mendu ML, Erickson KF, Hostetter TH, Winkelmayer WC, Olan G, Meyer RN, Hakim R, Sedor JR. Federal Funding for Kidney Disease Research: A Missed Opportunity. Am J Public Health. 2016 Mar;106(3):406-7. doi: 10.2105/AJPH.2015.303009. No abstract available. PMID 26885959
- [Background] System USRD. Annual Data Report 2015: Epidemiology of Kidney Disease in the United States. Washington DC: National Institutes of Health, National Institute of Diabetes and Digestive and Kidney Diseases; 2015
- [Background] Ojo A. Addressing the global burden of chronic kidney disease through clinical and translational research. Trans Am Clin Climatol Assoc. 2014;125:229-43; discussion 243-6. PMID 25125737
- [Background] Assari S. Distal, intermediate, and proximal mediators of racial disparities in renal disease mortality in the United States. J Nephropathol. 2016 Jan;5(1):51-9. doi: 10.15171/jnp.2016.09. Epub 2015 Dec 4. PMID 27047811
- [Background] Hsu CY, Lin F, Vittinghoff E, Shlipak MG. Racial differences in the progression from chronic renal insufficiency to end-stage renal disease in the United States. J Am Soc Nephrol. 2003 Nov;14(11):2902-7. doi: 10.1097/01.asn.0000091586.46532.b4. PMID 14569100
- [Background] Genovese G, Friedman DJ, Ross MD, Lecordier L, Uzureau P, Freedman BI, Bowden DW, Langefeld CD, Oleksyk TK, Uscinski Knob AL, Bernhardy AJ, Hicks PJ, Nelson GW, Vanhollebeke B, Winkler CA, Kopp JB, Pays E, Pollak MR. Association of trypanolytic ApoL1 variants with kidney disease in African Americans. Science. 2010 Aug 13;329(5993):841-5. doi: 10.1126/science.1193032. Epub 2010 Jul 15. PMID 20647424
- [Background] Freedman BI, Skorecki K. Gene-gene and gene-environment interactions in apolipoprotein L1 gene-associated nephropathy. Clin J Am Soc Nephrol. 2014 Nov 7;9(11):2006-13. doi: 10.2215/CJN.01330214. Epub 2014 Jun 5. PMID 24903390
- [Background] Parsa A, Kao WH, Xie D, Astor BC, Li M, Hsu CY, Feldman HI, Parekh RS, Kusek JW, Greene TH, Fink JC, Anderson AH, Choi MJ, Wright JT Jr, Lash JP, Freedman BI, Ojo A, Winkler CA, Raj DS, Kopp JB, He J, Jensvold NG, Tao K, Lipkowitz MS, Appel LJ; AASK Study Investigators; CRIC Study Investigators. APOL1 risk variants, race, and progression of chronic kidney disease. N Engl J Med. 2013 Dec 5;369(23):2183-96. doi: 10.1056/NEJMoa1310345. Epub 2013 Nov 9. PMID 24206458
- [Background] Goraya N, Simoni J, Jo C, Wesson DE. Dietary acid reduction with fruits and vegetables or bicarbonate attenuates kidney injury in patients with a moderately reduced glomerular filtration rate due to hypertensive nephropathy. Kidney Int. 2012 Jan;81(1):86-93. doi: 10.1038/ki.2011.313. Epub 2011 Aug 31. PMID 21881553
- [Background] Goraya N, Simoni J, Jo CH, Wesson DE. A comparison of treating metabolic acidosis in CKD stage 4 hypertensive kidney disease with fruits and vegetables or sodium bicarbonate. Clin J Am Soc Nephrol. 2013 Mar;8(3):371-81. doi: 10.2215/CJN.02430312. Epub 2013 Feb 7. PMID 23393104
- [Background] Goraya N, Simoni J, Jo CH, Wesson DE. Treatment of metabolic acidosis in patients with stage 3 chronic kidney disease with fruits and vegetables or oral bicarbonate reduces urine angiotensinogen and preserves glomerular filtration rate. Kidney Int. 2014 Nov;86(5):1031-8. doi: 10.1038/ki.2014.83. Epub 2014 Apr 2. PMID 24694986
- [Background] Navaneethan SD, Schold JD, Arrigain S, Jolly SE, Nally JV Jr. Cause-Specific Deaths in Non-Dialysis-Dependent CKD. J Am Soc Nephrol. 2015 Oct;26(10):2512-20. doi: 10.1681/ASN.2014101034. Epub 2015 Jun 4. PMID 26045089
- [Background] Honeycutt AA, Segel JE, Zhuo X, Hoerger TJ, Imai K, Williams D. Medical costs of CKD in the Medicare population. J Am Soc Nephrol. 2013 Sep;24(9):1478-83. doi: 10.1681/ASN.2012040392. Epub 2013 Aug 1. PMID 23907508
- [Background] Banks J, Marmot M, Oldfield Z, Smith JP. Disease and disadvantage in the United States and in England. JAMA. 2006 May 3;295(17):2037-45. doi: 10.1001/jama.295.17.2037. PMID 16670412
- [Background] So BH, Methven S, Hair MD, Jardine AG, MacGregor MS. Socio-economic status influences chronic kidney disease prevalence in primary care: a community-based cross-sectional analysis. Nephrol Dial Transplant. 2015 Jun;30(6):1010-7. doi: 10.1093/ndt/gfu408. Epub 2015 Jan 13. PMID 25586406
- [Background] Vart P, Gansevoort RT, Coresh J, Reijneveld SA, Bultmann U. Socioeconomic measures and CKD in the United States and The Netherlands. Clin J Am Soc Nephrol. 2013 Oct;8(10):1685-93. doi: 10.2215/CJN.12521212. Epub 2013 Jun 27. PMID 23813554
- [Background] Vart P, Reijneveld SA, Bultmann U, Gansevoort RT. Added value of screening for CKD among the elderly or persons with low socioeconomic status. Clin J Am Soc Nephrol. 2015 Apr 7;10(4):562-70. doi: 10.2215/CJN.09030914. Epub 2015 Mar 16. PMID 25779994
- [Background] Kurella-Tamura M, Goldstein BA, Hall YN, Mitani AA, Winkelmayer WC. State medicaid coverage, ESRD incidence, and access to care. J Am Soc Nephrol. 2014 Jun;25(6):1321-9. doi: 10.1681/ASN.2013060658. Epub 2014 Mar 20. PMID 24652791
- [Background] Kangovi S, Barg FK, Carter T, Long JA, Shannon R, Grande D. Understanding why patients of low socioeconomic status prefer hospitals over ambulatory care. Health Aff (Millwood). 2013 Jul;32(7):1196-203. doi: 10.1377/hlthaff.2012.0825. PMID 23836734
- [Background] Hoy WE, Wang Z, Baker PR, Kelly AM. Reduction in natural death and renal failure from a systematic screening and treatment program in an Australian Aboriginal community. Kidney Int Suppl. 2003 Feb;(83):S66-73. doi: 10.1046/j.1523-1755.63.s83.14.x. PMID 12864878
- [Background] Record NB, Onion DK, Prior RE, Dixon DC, Record SS, Fowler FL, Cayer GR, Amos CI, Pearson TA. Community-wide cardiovascular disease prevention programs and health outcomes in a rural county, 1970-2010. JAMA. 2015 Jan 13;313(2):147-55. doi: 10.1001/jama.2014.16969. PMID 25585326
- [Background] McClure JB. Are biomarkers useful treatment aids for promoting health behavior change? An empirical review. Am J Prev Med. 2002 Apr;22(3):200-7. doi: 10.1016/s0749-3797(01)00425-1. PMID 11897465
- [Background] Crews DC, Boulware LE, Gansevoort RT, Jaar BG. Albuminuria: is it time to screen the general population? Adv Chronic Kidney Dis. 2011 Jul;18(4):249-57. doi: 10.1053/j.ackd.2011.06.004. PMID 21782131
- [Background] Hoerger TJ, Wittenborn JS, Zhuo X, Pavkov ME, Burrows NR, Eggers P, Jordan R, Saydah S, Williams DE. Cost-effectiveness of screening for microalbuminuria among African Americans. J Am Soc Nephrol. 2012 Dec;23(12):2035-41. doi: 10.1681/ASN.2012040347. PMID 23204444
- [Background] Tuot DS, Peralta CA. To screen or not to screen: that is not (yet) the question. Clin J Am Soc Nephrol. 2015 Apr 7;10(4):541-3. doi: 10.2215/CJN.02150215. Epub 2015 Mar 16. No abstract available. PMID 25779993
- [Background] Vargas RB, Norris KC. Kidney disease progression and screening cost-effectiveness among African Americans. J Am Soc Nephrol. 2012 Dec;23(12):1915-6. doi: 10.1681/ASN.2012101028. Epub 2012 Nov 15. No abstract available. PMID 23160510
- [Background] Maziarz M, Black RA, Fong CT, Himmelfarb J, Chertow GM, Hall YN. Evaluating risk of ESRD in the urban poor. J Am Soc Nephrol. 2015 Jun;26(6):1434-42. doi: 10.1681/ASN.2014060546. Epub 2014 Dec 4. PMID 25475746
- [Background] Wilson DK, Kitzman-Ulrich H, Resnicow K, Van Horn ML, St George SM, Siceloff ER, Alia KA, McDaniel T, Heatley V, Huffman L, Coulon S, Prinz R. An overview of the Families Improving Together (FIT) for weight loss randomized controlled trial in African American families. Contemp Clin Trials. 2015 May;42:145-57. doi: 10.1016/j.cct.2015.03.009. Epub 2015 Mar 30. PMID 25835731
- [Background] Wilson DK, Kitzman-Ulrich H, Williams JE, Saunders R, Griffin S, Pate R, Van Horn ML, Evans A, Hutto B, Addy CL, Mixon G, Sisson SB. An overview of "The Active by Choice Today" (ACT) trial for increasing physical activity. Contemp Clin Trials. 2008 Jan;29(1):21-31. doi: 10.1016/j.cct.2007.07.001. Epub 2007 Jul 17. PMID 17716952
- [Background] Wilson DK, Trumpeter NN, St George SM, Coulon SM, Griffin S, Lee Van Horn M, Lawman HG, Wandersman A, Egan B, Forthofer M, Goodlett BD, Kitzman-Ulrich H, Gadson B. An overview of the "Positive Action for Today's Health" (PATH) trial for increasing walking in low income, ethnic minority communities. Contemp Clin Trials. 2010 Nov;31(6):624-33. doi: 10.1016/j.cct.2010.08.009. Epub 2010 Aug 27. PMID 20801233
- [Background] Kitzman H, Dodgen L, Mamun A, Slater JL, King G, Slater D, King A, Mandapati S, DeHaven M. Community-based participatory research to design a faith-enhanced diabetes prevention program: The Better Me Within randomized trial. Contemp Clin Trials. 2017 Nov;62:77-90. doi: 10.1016/j.cct.2017.08.003. Epub 2017 Aug 12. PMID 28807739
- [Background] Bibbins-Domingo K, Chertow GM, Fried LF, Odden MC, Newman AB, Kritchevsky SB, Harris TB, Satterfield S, Cummings SR, Shlipak MG. Renal function and heart failure risk in older black and white individuals: the Health, Aging, and Body Composition Study. Arch Intern Med. 2006 Jul 10;166(13):1396-402. doi: 10.1001/archinte.166.13.1396. PMID 16832005
- [Background] Bibbins-Domingo K, Pletcher MJ, Lin F, Vittinghoff E, Gardin JM, Arynchyn A, Lewis CE, Williams OD, Hulley SB. Racial differences in incident heart failure among young adults. N Engl J Med. 2009 Mar 19;360(12):1179-90. doi: 10.1056/NEJMoa0807265. PMID 19297571
- [Background] Gillespie BW, Morgenstern H, Hedgeman E, Tilea A, Scholz N, Shearon T, Burrows NR, Shahinian VB, Yee J, Plantinga L, Powe NR, McClellan W, Robinson B, Williams DE, Saran R. Nephrology care prior to end-stage renal disease and outcomes among new ESRD patients in the USA. Clin Kidney J. 2015 Dec;8(6):772-80. doi: 10.1093/ckj/sfv103. Epub 2015 Nov 3. PMID 26613038
- [Background] Bauer UE, Briss PA, Goodman RA, Bowman BA. Prevention of chronic disease in the 21st century: elimination of the leading preventable causes of premature death and disability in the USA. Lancet. 2014 Jul 5;384(9937):45-52. doi: 10.1016/S0140-6736(14)60648-6. Epub 2014 Jul 1. PMID 24996589
- [Background] Jenkins DJA, Boucher BA, Ashbury FD, Sloan M, Brown P, El-Sohemy A, Hanley AJ, Willett W, Paquette M, de Souza RJ, Ireland C, Kwan N, Jenkins A, Pichika SC, Kreiger N. Effect of Current Dietary Recommendations on Weight Loss and Cardiovascular Risk Factors. J Am Coll Cardiol. 2017 Mar 7;69(9):1103-1112. doi: 10.1016/j.jacc.2016.10.089. PMID 28254171
- [Background] Thomson CA, Ravia J. A systematic review of behavioral interventions to promote intake of fruit and vegetables. J Am Diet Assoc. 2011 Oct;111(10):1523-35. doi: 10.1016/j.jada.2011.07.013. PMID 21963019
- [Background] Sharan AD, Schroeder GD, West ME, Vaccaro AR. Understanding a Value Chain in Health Care. J Spinal Disord Tech. 2015 Oct;28(8):291-3. doi: 10.1097/BSD.0000000000000319. PMID 26356585
- [Background] Mundt L, Shanahan K. Textbook of Urinalysis and Body Fluids. 2nd ed. Philadelphia, PA: Lippincott Williams & Wilkins; 2011.
- [Background] Ozyilmaz A, de Jong PE, Bakker SJL, Visser ST, Thio C, Gansevoort RT; PREVEND Study Group. Screening for elevated albuminuria and subsequently hypertension identifies subjects in which treatment may be warranted to prevent renal function decline. Nephrol Dial Transplant. 2017 Apr 1;32(suppl_2):ii200-ii208. doi: 10.1093/ndt/gfw414. PMID 28031343
- [Background] Carrero JJ, Grams ME, Sang Y, Arnlov J, Gasparini A, Matsushita K, Qureshi AR, Evans M, Barany P, Lindholm B, Ballew SH, Levey AS, Gansevoort RT, Elinder CG, Coresh J. Albuminuria changes are associated with subsequent risk of end-stage renal disease and mortality. Kidney Int. 2017 Jan;91(1):244-251. doi: 10.1016/j.kint.2016.09.037. Epub 2016 Dec 4. PMID 27927597
- [Background] Levey AS, Becker C, Inker LA. Glomerular filtration rate and albuminuria for detection and staging of acute and chronic kidney disease in adults: a systematic review. JAMA. 2015 Feb 24;313(8):837-46. doi: 10.1001/jama.2015.0602. PMID 25710660
- [Background] Deci EL, Eghrari H, Patrick BC, Leone DR. Facilitating internalization: the self-determination theory perspective. J Pers. 1994 Mar;62(1):119-42. doi: 10.1111/j.1467-6494.1994.tb00797.x. PMID 8169757
- [Background] Carithers TC, Talegawkar SA, Rowser ML, Henry OR, Dubbert PM, Bogle ML, Taylor HA Jr, Tucker KL. Validity and calibration of food frequency questionnaires used with African-American adults in the Jackson Heart Study. J Am Diet Assoc. 2009 Jul;109(7):1184-1193. doi: 10.1016/j.jada.2009.04.005. PMID 19559135
- [Background] Subar AF. Developing dietary assessment tools. J Am Diet Assoc. 2004 May;104(5):769-70. doi: 10.1016/j.jada.2004.02.007. No abstract available. PMID 15127062
- [Derived] Kitzman H, Montgomery AH, Khan M, Mamun A, Tecson KM, Allison P, Simoni J, Wesson DE. The Fruit and Veggies for Kidney Health Study: A Prospective Randomized Trial. Kidney Med. 2023 Oct 23;5(12):100736. doi: 10.1016/j.xkme.2023.100736. eCollection 2023 Dec. PMID 38046912

DOCUMENTS (1):
  • Informed Consent Form (2019-01-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT03832166/ICF_000.pdf